CLINICAL TRIAL: NCT00150228
Title: A Twelve-Week Double-Blind, Placebo-Controlled, Randomized, Multicenter Study Evaluating the Safety and Efficacy of a Flexible-Dosing Strategy for CP-526,555 ( 0.5 mg to 2.0 mg Total Daily Dose ) in Smoking Cessation
Brief Title: 12 Week Evaluation of the Safety and Efficacy of a Flexible Dose of CP-526,555 and Placebo for Smoking Cessation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3051016
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2007-06-04 (Estimated); Status verified 2007-05

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

INTERVENTIONS:
Drug: CP-526,555 (varenicline)

SUMMARY:
The purpose of the study was to measure the safety and efficacy of a 12-week flexible dosing strategy of CP-526,555 compared with placebo for smoking cessation. Post-treatment follow-up of smoking status to one year from randomization was performed in a non-treatment extension Protocol A3051019

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have smoked an average of at least ten cigarettes per day during the past year
* No period of abstinence greater than three months in the past year

Exclusion Criteria:

* Subjects with history of clinically significant cardiovascular disease
* Subjects with uncontrolled hypertension.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2001-12; Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
4-week continuous quit rate (CQR) at Weeks 4-7 and 9-12 .

SECONDARY OUTCOMES:
Continuous abstinence rate from target quit date to end of treatment (Week 12)
7-day point prevalence of abstinence at Week 12
Number of cigarettes smoked per day
Urge to smoke and withdrawal symptoms assessed by Minnesota Nicotine Withdrawal Scale
Rewarding effects of smoking assessed by Smoking Effects Inventory
weight change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (7):
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Albert Lea, Minnesota
  - Pfizer Investigational Site, Rochester, Minnesota
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Providence, Rhode Island
  - Pfizer Investigational Site, La Crosse, Wisconsin
  - Pfizer Investigational Site, Madison, Wisconsin

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Niaura R, Hays JT, Jorenby DE, Leone FT, Pappas JE, Reeves KR, Williams KE, Billing CB Jr. The efficacy and safety of varenicline for smoking cessation using a flexible dosing strategy in adult smokers: a randomized controlled trial. Curr Med Res Opin. 2008 Jul;24(7):1931-41. doi: 10.1185/03007990802177523. Epub 2008 May 29. PMID 18513462
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051016&StudyName=+12+Week+Evaluation+of+the+Safety+and+Efficacy+of+a+Flexible+Dose+of+CP%2D526%2C555+and+Placebo+for+Smoking+Cessation